CLINICAL TRIAL: NCT04689204
Title: A Study of CTA30X Cell Injection in the Treatment of Relapsed or Refractory CD19-positive B-line Hematological Malignancies
Brief Title: A Study of CTA30X Cell Injection in Patients With Relapsed or Refractory CD19-positive B-line Hematological Malignancies
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: He Huang (Other)
Collaborators: Nanjing Bioheng Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, He Huang, Clinical Professor, Zhejiang University
Organization: Zhejiang University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BHCT-CTA30X-01
Record Dates: First submitted 2020-12-25; First posted 2020-12-30 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Acute Lymphoblastic Leukemia; Non-hodgkin Lymphoma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Administration of CTA30X (Experimental): Dose escalation follows the standard 3+3 dose escalation design. A total of 3 dose levels are set for subjects.
  Interventions: Drug: CTA30X

INTERVENTIONS:
Drug: CTA30X — CTA30X cell injection by intravenous infusion
  Other Names: CTA30X cell injection

SUMMARY:
A study of CTA30X cell injection in the treatment of relapsed or refractory CD19-positive B-line hematological malignancies

DETAILED DESCRIPTION:
This is a single arm, open-label, single-center study. This study is indicated for relapsed or refractory CD19+ B-line hematological malignancy: B-ALL and B-NHL. the selection of dose levels and the number of subjects are based on clinical tiral of similar foreign products. 3 groups of patients will be enrolled, 36 in each group. Primary objective is to explore the safety, main consideration is dose-related safety.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria applicable to ALL only:

1. Male or female aged ≥ 3 and <70 years old;
2. Histologically confirmed diagnosis of CD19+ B-ALL per the US National Comprehensive Cancer Network (NCCN) Clinical Practice Guidelines for Acute Lymphoblastic Leukemia (2016.v1);
3. Relapsed or refractory CD19+ B-ALL (meeting one of the following conditions):

   1. CR not achieved after standardized chemotherapy;
   2. CR achieved following the first induction, but CR duration is ≤ 12 months;
   3. Ineffective after first or multiple remedial treatments;
   4. 2 or more recurrences;
4. The number of primordial cells (lymphoblast and prolymphocyte) in bone marrow is >5% (morphology) and/or >1% (Flow cytometry);
5. Philadelphia-chromosome-negative (Ph-) patients; or Philadelphiachromosome-positive (Ph+) patients who cannot tolerate TKI treatments or do not respond to 2 TKI treatments;

Inclusion criteria applicable to NHL only:

1. Male or female aged ≥ 18 and <70 years old;
2. Histologically confirmed diagnosis per WHO Classification Criteria for Lymphocytic Tumors 2016, including DLBCL(NOS), follicular lymphoma, Chronic lymphoblastic leukemia/small lymphoblastic lymphoma transforms DLBCL, PMBCL and high grade B cell lymphoma;
3. Relapsed or refractory DLBCL (meeting one of the following conditions):

   1. No remission or recurrence after receiving second-line or above chemotherapy;
   2. Primary drug resistance;
   3. Recurrence after autologous hematopoietic stem cell transplantation

Applicable standards for ALL and NHL:

1. Total bilirubin ≤ 51umol/L, ALT and AST ≤ 3 times of upper limit of normal, creatinine ≤ 176.8umol/L;
2. Echocardiogram shows left ventricular ejection fraction (LVEF) ≥ 50%;
3. No active infection in the lungs, blood oxygen saturation by sucking air is ≥92%;
4. Estimated survival time ≥ 3 months;
5. ECOG performance status 0 to 2;

Exclusion Criteria:

1. Patients with extramedullary lesions, except those with CNSL (CNS-1) under effective control (for ALL patients only);
2. Confirmed diagnosis of lymphoblastic crisis of chronic myeloid leukemia, Burkitt's leukemia/lymphoma per WHO Classification Criteria (for ALL patients only);
3. Patients with hereditary syndrome such as Fanconi anemia, Kostmann syndrome, Shwachman syndrome or any other known bone marrow failure syndrome (for ALL patients only);
4. Patients with intracranial extralateral lesions (cerebrospinal fluid tumor cells and/or intracranial lymphoma invasion shown by MRI) (for NHL patients only);
5. Extensive involvement of gastrointestinal lymphoma (for NHL patients only);
6. Radiotherapy, chemotherapy and monoclonal antibody within 1 week before screening;
7. Have a history of allergy to any of the components in the cell products;
8. Prior treatment with any CAR T cell product or other genetically-modified T cell therapies;
9. According to the New York heart association (NYHA) cardiac function classification criteria, Subjects with grade III or IV cardiac insufficiency;
10. Myocardial infarction, cardioangioplasty or stenting, unstable angina pectoris, or other severe cardiac diseases within 12 months of enrollment;
11. Severe primary or secondary hypertension of grade 3 or above (WHO Hypertension Guidelines, 1999);
12. Electrocardiogram shows prolonged QT interval, severe heart diseases such as severe arrhythmia in the past;
13. History of craniocerebral trauma, conscious disturbance, epilepsy, cerebrovascular ischemia, and cerebrovascular hemorrhagic diseases;
14. Patients with severe active infections (excluding simple urinary tract infection and bacterial pharyngitis).
15. History of other primary cancer, except for the following conditions:

    1. Cured non-melanoma after resection, such as basal cell carcinoma of the skin;
    2. Cervical cancer in situ, localized prostate cancer, ductal cancer in situ with disease-free survival ≥ 2 years after adequate treatment;
16. Patients with autoimmune diseases requiring treatment, patients with immunodeficiency or requiring immunosuppressive therapy;
17. Patients with graft-versus-host disease (GVHD);
18. If HBsAg positive at screening, HBV DNA copy number detected by PCR in patients with active hepatitis B > 1000 (if HBV DNA copy number≤1000, routine antiviral therapy is required after enrollment), as well as CMV, hepatitis C, syphilis infection;
19. Patients who have participated in any other clinical studies within 2 weeks prior to screening;
20. Pregnant and breast-feeding women and the subjects who are fertile and unable to take effective contraceptive measures (regardless of the gender);
21. Any situations that the investigator believes may increase the risk of patients or interfere with the results of study.

Ages: 3 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-12-29 (Actual); Primary Completion 2022-12-29 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Baseline up to 28 days after CTA30X infusion
  Adverse events assessed according to NCI-CTCAE v5.0 criteria
Incidence of treatment-emergent adverse events (TEAEs) | Up to 2 years after CTA30X infusion
  Incidence of treatment-emergent adverse events [Safety and Tolerability]

SECONDARY OUTCOMES:
B-cell acute lymphocytic leukemia (B-ALL), Overall response rate (ORR) | Month 1 and 3
  Assessment of ORR (ORR = CR + CRi ) at Month 1 and 3
B-ALL, MRD negative overall response rate (MRD- ORR) | 3 months
  Assessment of MRD negative overall response rate (MRD- ORR) at 3 months after CTA30X infusion
B-ALL, ORR | Month 6, 12, 18 and 24
  Assessment of ORR at Month 6, 12, 18 and 24
B-ALL, Event-free survival (EFS) | Month 6, 12, 18 and 24
  From the first infusion of CTA30X to the occurrence of any event, including death, relapse or gene relapse, disease progression (any one occurs first), and the last visit
B cell non-hodgkin's lymphoma (B-NHL), Overall response rate (ORR) | weeks 4, 12, months 6, 12, 18 and 24
  Assessment of ORR (ORR = CR + PR ) per Lugano 2014 criteria

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital，College of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No